CLINICAL TRIAL: NCT06135831
Title: Effect of the Consumption of Vitamin C, D3, Ca Supplements and Olive Paste Enriched With Mountain Tea on Bone Metabolism Indices in Postmenopausal Women With Increased Osteoporosis' Risk: A Prospective Interventional Study
Brief Title: Effect of Consumption of Supplements and Enriched Olive Paste on Bone Metabolism Indices
Acronym: Osteoporosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Aegean (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Osteo21
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Osteopenia or Osteoporosis
Keywords: postmenopausal; osteopenia; osteoporosis; supplements; functional olive paste
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis | interventions — Ascorbic Acid; Fumigant 93; Calcium; Magnesium; Diphosphonates; Vitamin D

STUDY DESIGN:
Intervention Model Description: Each study arm received different supplementation.
Who Masked: Participant
Masking Description: It was a single blinded nutritional intervention, where only participants didn't know in which group was recruited.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Calciovitmag (CDCaMg) (Experimental): Daily supplementation of diet with vitamin C (1000 mg), vitamin D3 (500 mg), calcium (Ca) (500 mg ) and magnesium (Mg) (300 mg)
  Interventions: Other: Calciovitmag (CDCaMg)
- Control (Placebo Comparator): Daily supplementation of diet with vitamin D3 (500 mg), Ca (500 mg) and Mg (300 mg)
  Interventions: Other: Control
- Phosphorovitmag (PDCaMg) (Experimental): Daily supplementation of diet with bisphosphonates (150 mg), vitamin D3 (500 mg), Ca (500 mg ) and Mg (300 mg)
  Interventions: Other: Phosporovitmag (PDCaMg)
- Functional Olive paste (Experimental): Daily supplementation of diet with 364 mg polyphenols via 50 g of an innovative functional food (Kalamata olive paste with mountain tea rich in polyphenols, (total phenolics 7,28±3.11 gallic acid/g) along with vitamin D3 (500 mg), Ca (500 mg) and Mg (300 mg)
  Interventions: Other: Functional olive paste

INTERVENTIONS:
Other: Functional olive paste — Homogenised olive pastes, enriched with mountain tea, were supplied by two ac-credited Greek olive oil and olive products companies, Arcadian Taste and GAEA. The fortified olive pastes, contained 7.5 g of extra virgin olive oil, 3.75 g of salt, 3.75 g of grated oregano, 3.75 g of grated pepper, 7.5 g of grated garlic, 6.25 g of orange juice, 65 g of Kala-mon olives without seeds and 3 g of mountain tea and weighted 100 gr per portion size, as well.
  Other Names: Olive paste enriched with mountain tea
  Arms: Functional Olive paste
Other: Calciovitmag (CDCaMg) — Vitamin C (1000 mg), vitamin D3 (500 mg), Calcium (Ca) (500 mg ) and Magnesium (Mg) (300 mg)/day
  Other Names: Vitamin C and D, Calcium and Magnesium
  Arms: Calciovitmag (CDCaMg)
Other: Phosporovitmag (PDCaMg) — Bisphosphonates (150 mg), vitamin D3 (500 mg), Ca (500 mg ) and Mg (300 mg)/daily
  Other Names: Bisphosphonates, Vitamin D, Calcium and Magnesium
  Arms: Phosphorovitmag (PDCaMg)
Other: Control — Vitamin D3 (500 mg), Calcium (500 mg) and Magnesium (300 mg)/daily
  Arms: Control

SUMMARY:
It was a prospective randomized controlled trial. A sample of 115 apparently healthy post-menopausal women(45 -75 years of age) randomized into four groups and received supplements of Ca, Vitamin D and Mg with or without enriched olive paste and with or without Vitamin C. Changes in calciregulatory hormone were evaluated at the beginning of the study, at 5 and 12 months . Blood levels of vitamin D, vitamin C, Ca, Mg, the lipid profile, anthropometric indices and bone density were assessed at the beginning and at the end of the study.

DETAILED DESCRIPTION:
: It was a prospective randomized controlled trial. A sample of 115 apparently healthy post-menopausal women(45 -75 years of age) randomized into four groups: (I) nutritional intervention group(n=40) received daily 1000mg vitamin C, 500mg vitamin D3, 500mg calcium(Ca) and 300mg magnesium (Mg); (II) control group(n=42) received daily 500mg vitamin D3, 500mg Ca and 300mg Mg; (III) nutritional intervention group (n=18) received daily 150mg bisphosphonates, 500mg vitamin D3, 500mg Ca and 300mg Mg; and (IV) nutritional intervention group (n=15) received daily about 364 mg polyphenols via an innovative functional food (50g olive paste enriched with mountain tea extract) along with 500mg vitamin D3, 500mg Ca and 300mg Mg. Groups I -III received supplementation for a year whereas group IV for 5 months. Changes in calciregulatory hormone parathormone (PTH) were evaluated at the beginning of the study as well as at 5 and 12 months intervals. Blood levels of vitamin D, vitamin C, Ca, Mg and the lipid profile were assessed at the beginning and at the end of the study. Anthropometric indices (weight, body fat(Kg), Body Mass Index(BMI) and bone mineral density(BMD) were evaluated at the beginning and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 45 to 75 years old
* Screening for osteoporosis (t-score ≤ - 1 normal bone density, t-score ≤ 2.5 osteoporosis ) and osteopenia of the femur strength or spine (t-score between -1 and -2.5 )

Exclusion Criteria:

* Age > 75 y.o. and <45 y.o
* Diagnosed with chronic diseases including cancer, diabetes, coronary heart disease and stroke

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only postmenopausal women with osteopenia or osteoporosis were eligible for participation
Enrollment: 115 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in calciregulatory hormone parathormone | 12 months
  Changes in calciregulatory hormone parathormone (PTH) at baseline, 5 and 12 months

SECONDARY OUTCOMES:
Changes in Vitamin D | 12 months
  Changes in Vitamin D at baseline and 12 months
Changes in Calcium | 12 months
  Changes in Calcium at baseline and 12 months
Changes in Vitamin C | 12 months
  Changes in Vitamin C at baseline and 12 months
Changes in Magnesium | 12 months
  Changes in Magnesium at baseline and 12 months
Changes in serum lipids | 12 months
  Changes in serum lipids at baseline and 12 months
Changes in body weight, body mass index and body fat | 12 months
  Changes in body weight, body mass index and body fat at baseline and 12 months
Changes in Bone Mineral Density | 12 months
  Changes in Bone Mineral Density at baseline and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of the Aegean, Myrina, Limnos/Lesvos, Greece

IPD SHARING:
Plan to Share IPD: No
No one individual participant data will be shared